CLINICAL TRIAL: NCT06310278
Title: Ossiview Normative Mobility Data Collection Protocol
Status: Recruiting | Type: Observational
Sponsor: Audioptics Medical Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 1030312
Record Dates: First submitted 2024-03-02; First posted 2024-03-15 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Conductive Hearing Loss, Middle Ear
Keywords: optical coherence tomography
MeSH Terms: conditions — Hearing Loss, Conductive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normal-hearing
  Interventions: Diagnostic Test: Ossicular mobility measurement

INTERVENTIONS:
Diagnostic Test: Ossicular mobility measurement — Measurements of ossicular mobility i.e. the dynamic velocity of middle ear structures (umbo of malleus and incus at the incudostapedial joint) normalized to sound pressure incident on the tympanic membrane.

SUMMARY:
The goal of this observational study is to learn about the sound-induced vibration level of certain structures in the middle ear in the normal-hearing population. The targeted structures are part of a chain of structures responsible for conducting sound within the auditory system and so their ability to vibrate normally in response to sound is relevant to the diagnosis of conductive hearing loss.

The main questions the study aims to answer are:

* What are the mean and variance of the normal sound-induced vibration level at two anatomical locations, the umbo of the malleus and the tip of the incus?
* Are there any significant differences in these vibrational responses associated with sex or age?

Participants will have their ossicular mobility measured with an investigational medical device that sends light into the middle ear and measures the motion-induced phase shift on light reflected from the target structures when a sound stimulus is presented. Standard hearing tests including audiometry and tympanometry will also be performed to confirm the normal hearing status of participants.

ELIGIBILITY:
Inclusion Criteria:

* Normal-hearing
* Over the age of 18
* At least one of incus or umbo visible under otoscopic examination
* Type A 226Hz tympanogram with peak static compliance occurring at pressure between -99mmH20 and +50mmH20 and peak static compliance in the range from 0.3 to 1.6 cc

Exclusion Criteria:

* Audiometric air conduction thresholds greater than 40 dBHL at 500 Hz, 750 Hz, 1000 Hz, 1500Hz, 2000 Hz, 3000 Hz
* Audiometric air bone gap greater than 5dB at 500Hz, 750Hz, 1000Hz, 1500Hz, 2000Hz and 3000Hz
* Self-reported history of ear infection in the previous 3 months
* Self-reported history of middle ear surgery in the last 5 years
* Self-reported history of tympanic membrane perforation within the last 5 years
* Self-reported medical treatment for any ear-related disorder within the last 5 years
* Evidence of perforation, tympanosclerosis, otitis externa, thickened or fibrotic eardrum, mycosis, fluid, infection or other ear abnormality under otoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Minimum 120 normal-hearing subjects including at least 10 male and 10 female subjects in each age group 18-30, 30-40, 40-50, 50-60 and 60+
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Umbo mobility | At study completion (6 months)
  Estimated mean and variance of mobility in mm/s/Pa in the normal-hearing population measured at the umbo of the malleus at 500Hz, 750Hz, 1000Hz, 1500Hz, 2000Hz and 3000Hz stimulus frequencies.
Incus mobility | At study completion (6 months)
  Estimated mean and variance of mobility in mm/s/Pa in the normal-hearing population measured at the incus lateral to the incudostapedial joint at 500Hz, 750Hz, 1000Hz, 1500Hz, 2000Hz and 3000Hz stimulus frequencies.

SECONDARY OUTCOMES:
Dependence on age and sex | At study completion (6 months)
  p-values for dependence on age, sex and age-sex interaction at each stimulus frequency within two-way ANOVA.

CONTACTS AND LOCATIONS:
Overall Officials: David P Morris, FRCS(Oto), Principal Investigator — Nova Scotia Health
Locations (1):
- Audioptics Medical, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No